CLINICAL TRIAL: NCT02165475
Title: Combination Therapy With Biofeedback, Loperamide and Stool Bulking Agents is Effective for the Treatment of Fecal Incontinence in Women - a Randomized Controlled Trial
Brief Title: Combination Therapy With Biofeedback, Loperamide and Stool Bulking Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Jenny Sjödahl, PhD, University Hospital, Linkoeping
Purpose: Treatment
Other Study IDs: Dnr 02-220
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- medical treatment (Experimental)
  Interventions: Drug: Loperamide; Drug: Stool bulking agent (stericulia or isphagula husk)
- combination of the two treatments (Experimental)
  Interventions: Other: Combination of biofeedback and medical treatment

INTERVENTIONS:
Behavioral: Biofeedback
  Arms: Biofeedback
Drug: Loperamide
  Arms: medical treatment
Drug: Stool bulking agent (stericulia or isphagula husk)
  Arms: medical treatment
Other: Combination of biofeedback and medical treatment
  Arms: combination of the two treatments

SUMMARY:
Background: Biofeedback and medical treatments have been extensively used for moderate fecal incontinence. There is limited data comparing and combining these two treatments.

Aim: To evaluate the effect of biofeedback and medical treatments, separately and in combination.

Methods: Sixty-five consecutive female patients, referred to a tertial center for fecal incontinence were included. The patients were randomized to start with either biofeedback (4-6 months) or medical treatment with loperamide and stool-bulking agents (2 months). Both groups continued with a combination treatments, i.e. medical treatment was added to biofeedback and vice versa. A two-week prospective bowel symptom diary and anorectal physiology were evaluated at baseline, after single- and combination treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients with at least one or more episodes of FI during a period of 2 weeks as recorded by bowel function diary
* Patients from whom written consent was obtained

Exclusion Criteria:

* Previous congenital or acquired spinal injury, spinal tumour or spinal surgery
* Presence of neurological diseases or peripheral vascular disease
* Uncontrolled diabetes mellitus
* Congenital anorectal malformations
* Recent colorectal or gastrointestinal surgery
* Presence of external full-thickness rectal prolapse
* Inflammatory bowel disease
* Chronic diarrhoea
* Use of tibial nerve or sacral nerve stimulations
* Ongoing pregnancy
* Any malignant disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
symptom diary | Up to eight months

CONTACTS AND LOCATIONS:
Locations (1):
- Pelvic floor unit, University hospital of Linköping, Linköping, Sweden